CLINICAL TRIAL: NCT00830661
Title: A Randomized, Prospective, Multi-Centered Study Comparing Clinical Outcomes of the Ligation of Intersphincteric Fistula Tract (LIFT)Procedure Versus Use of Anal Fistula Plug (AFP)in the Surgical Repair of Trans-Sphincteric Anal Fistulae of Cryptoglandular Origin
Brief Title: Ligation of Intersphincteric Fistula Tract (LIFT) Procedure Versus Use of an Anal Fistula Plug for Anal Fistula Repair
Acronym: LIFT vs PLUG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Colon and Rectal Surgery Associates, Ltd. (Other)
Collaborators: University of Pennsylvania (Other); University of Ottawa (Other); Massachusetts General Hospital (Other)
Responsible Party: Dr. Stanley M. Goldberg, MD Study Director, University of Minnesota/Colon and Rectal Surgery Associates. Ltd
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMG1108
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Anal Fistula
Keywords: transsphincteric anal fistula; cryptoglandular origin; anal fistula repair; Ligation of Intersphincteric Fistula Track (LIFT) procedure; anal fistula plug (Plug); surgical repair
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LIFT (Active Comparator): those subjects receiving the Ligation of Intersphincteric Fistula Track procedure
  Interventions: Procedure: Ligation of intersphincteric fistula track procedure
- Plug (Active Comparator): those subjects randomized to the receive the placement of the porcine anal fistula plug
  Interventions: Procedure: anal fistula plug

INTERVENTIONS:
Procedure: Ligation of intersphincteric fistula track procedure — Subjects randomized to this arm will receive the ligation of the intersphincteric fistula track (LIFT) procedure. This procedure will be performed as per standard operating procedure.
  Arms: LIFT
Procedure: anal fistula plug — placement of the porcine anal fistula plug as per the instructions for use in product packaging
  Arms: Plug

SUMMARY:
Anal fistulae are a difficult problem to treat. The optimal treatment for fistula involving the anal sphincter is unclear. Two standardly used methods of treatment are the ligation of intersphincteric fistula track (LIFT) procedure and the use of an anal fistula plug. The purpose of this study is to exam the rate of fistula closure between the LIFT procedure and the use of a fistula plug

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 years of age or older.
* Able to understand and provide informed consent or have a legally authorized representative capable of providing consent.
* Has a documented diagnosis, confirmed by physical exam and/or endorectal ultrasound (if available), of a trans-sphincteric fistula tract determined to be of cryptoglandular origin (primary or recurrent).

Exclusion Criteria:

* History or suspicion of Inflammatory Bowel Disease (Crohn's or Ulcerative colitis).
* History of connective tissue disease.
* Rectovaginal fistula.
* Presence of horseshoe fistula.
* History of immunosuppression therapy/treatment within previous six months.
* Presents of a proximal diversion and refractory fistula.
* Any physical conditions, disease, or disorder that would exclude subject from being a candidate for elective surgery.
* Known history of allergy to pork or pork products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2009-03; Primary Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure of this study will be to compare the rate of fistula closure between the ligation of the intersphincteric fistula track (LIFT) procedure and the use of a porcine bioabsorbable anal fistula plug | 1month, 3 month, 6 month, 12 month postoperatively

SECONDARY OUTCOMES:
Secondary measures will include level of fecal incontinence, fecal incontinence quality of life, complication rates, and rate of closure after re-operation | 1 month, 3 month, 6 month, 12 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Heather L Rossi, MD, Principal Investigator — University of Minnesota/Colon and Rectal Surgery Associates, Ltd.; Husein Moloo, MD, Principal Investigator — University of Ottawa; Joshua Bleier, MD, Principal Investigator — University of Pennsylvania Health System; Liliana Bordeianou, MD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Colon and Rectal Surgery Associates, Ltd, Minneapolis, Minnesota
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
- University of Ottawa, Ottawa, Ontario, Canada